CLINICAL TRIAL: NCT02142816
Title: Non-invasive Assessment of Fluid Requirement During Surgery: a Comparison of Oesophageal Doppler and Pleth Variability Index
Brief Title: Fluid Requirement During Surgery PVI v Doppler
Acronym: PVIvDoppler
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YOR-A02089
Record Dates: First submitted 2014-05-15; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Colorectal Surgery; Major Abdominal Surgery
MeSH Terms: interventions — Echocardiography, Doppler

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doppler (Active Comparator): Fluid directed by oesophageal doppler
  Interventions: Device: Doppler
- PVI (Active Comparator): Fluid therapy directed by Pleth Variability Index
  Interventions: Other: PVI'

INTERVENTIONS:
Device: Doppler — Fluid therapy guided by doppler
  Arms: Doppler
Other: PVI' — Fluid therapy guided by PVI
  Arms: PVI

SUMMARY:
Targeting the amount of fluid given to measurements of the patients own fluid status during major abdominal surgery has been linked with improved speed of recovery of gut function and reduced length of hospital stay, mortality and complications.

Pleth variability index (PVI) offers a noninvasive, risk and pain free alternative to more invasive forms of monitoring to direct how much fluid to give.

The study aims primarily to measure and compare how much fluid is given when guided by PVI compared to the established technique; oesophageal doppler during major abdominal surgery.

The study will compare 40 patients undergoing major elective abdominal surgery. Patients will receive intraoperative fluid guided by either oesophageal doppler or PVI. Secondarily, the study will examine biochemical markers, length of hospital stay and how frequently complications occur

ELIGIBILITY:
Inclusion Criteria:

* Major abdominal surgery
* Anaerobic Threshold >11 ml O2/kg/min
* VE/VCO2 <34 OR
* Low risk according to Consultant anaesthetist

Exclusion Criteria:

* Patients age less than 18
* Patient refused consent
* Patient unable to give consent
* Patient has had <24hrs to consider the Patient information Sheet
* Contraindication to Doppler Probe being inserted
* Emergency Procedure
* Patient has a ASA Grade 5
* Patient is receiving dialysis treatment
* Patient has a known hypersensitivity to hydroxyethyl starch or gelatin solutions
* Patients with renal failure with oliguria or anuria - not related to hypovolaemia
* Patients with a previously diagnosed dysrhythmia
* Patients who weight >100kg

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Difference between fluid volumes administered in the intra-operative period | End of operation

SECONDARY OUTCOMES:
Difference in 24 hour fluid balance | 24 hours
Post-operative morbiditiy survey | 7 days
Biochemical Markers of Tissue Perfusion | 24 hours
  Lactate and Base Excess

CONTACTS AND LOCATIONS:
Overall Officials: David Yates, MB ChB, Principal Investigator — York Teaching Hospital
Locations (1):
- York Teaching Hospital, York, N Yorks, United Kingdom